CLINICAL TRIAL: NCT02867163
Title: Does the Intraoperative Administration of Tranexamic Acid (TXA) Increase the Incidence of Deep Venous Thrombosis in Total Knee Arthroplasty?
Brief Title: Tranexamic Acid and Blood Clots in Knee Surgery
Status: Completed | Type: Observational
Sponsor: University of New Mexico (Other)
Responsible Party: Principal Investigator, David Siegel, Assistant Professor, University of New Mexico
Other Study IDs: TXA in TKR
Record Dates: First submitted 2016-08-04; First posted 2016-08-15 (Estimated); Results first posted 2019-05-20 (Actual); Last update posted 2019-05-20 (Actual); Status verified 2019-02

CONDITIONS: Venous Thrombosis
MeSH Terms: conditions — Venous Thrombosis | interventions — Tranexamic Acid

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Knee replacement patients receiving TXA: Patients who receive tranexamic acid during total knee replacement surgery
  Interventions: Drug: Tranexamic Acid

INTERVENTIONS:
Drug: Tranexamic Acid — Intravenous or local administration of TXA, in any dosage
  Other Names: Lysteda; Cyklokapron

SUMMARY:
This is an observational trial to estimate the incidence of deep vein thrombosis (DVT) in total knee replacement patients who received an intraoperative dose of tranexamic acid.

DETAILED DESCRIPTION:
This study is anticipated to consist of 30 participants over 18 years of age scheduled for total knee arthroplasty at Sandoval Regional Medical Center with administered intraoperative tranexamic acid, who do not meet the exclusion criteria. The patients will be examined on postoperative day 1. Lower-extremity ultrasound will be used to screen for deep vein thrombosis (DVT). Incidence data for DVT will then be compared with the historical incidence rate at our institution for total knee arthroplasty without the use of tranexamic acid, which is approximately 12%. Patients found on screening to have deep vein thrombosis will be referred for appropriate care.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients scheduled for total knee arthroplasty at Sandoval Regional Medical Center with an intraoperative dose of tranexamic acid

Exclusion Criteria:

* Previous deep vein thrombosis or pulmonary embolism episode
* Known coronary artery disease or peripheral vascular disease
* Previously diagnosed hypercoagulable states (e.g. Leiden factor V, antiphospholipid antibody, protein C or S deficiency)
* Pregnancy
* Creatinine clearance less than 30 ml/min
* Non-fluency in English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients having total knee replacement at Sandoval Regional Medical Center in Rio Rancho, New Mexico, and who receive an intraoperative dose of tranexamic acid to control surgical bleeding
Sampling Method: Non-Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2017-11-08 (Actual); Study Completion 2017-11-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David Siegel, MD, Principal Investigator — University of New Mexico
Locations (1):
- Sandoval Regional Medical Center, Rio Rancho, New Mexico, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Knee Replacement Patients Receiving TXA
Started | 25
Completed | 25
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Knee Replacement Patients Receiving TXA
Number analyzed (Participants) | 25
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 25

OUTCOME MEASURES:

1. Primary Outcome: Deep Vein Thrombosis
Description: Incidence of deep vein thrombosis diagnosed by ultrasound scan on postoperative day 1
Time Frame: One day
Measure: Count of Participants; unit: Participants
Arm/Group | Knee Replacement Patients Receiving TXA
Number analyzed (Participants) | 25
Participants | 2

ADVERSE EVENTS:
Time Frame: 3 days
Arm/Group | Knee Replacement Patients Receiving TXA
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 0/25
Other Adverse Events (participants affected / at risk) | 0/25

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-08-03): https://cdn.clinicaltrials.gov/large-docs/63/NCT02867163/Prot_SAP_000.pdf